CLINICAL TRIAL: NCT01973348
Title: Comparison of AmblyzTM Glasses and Patching for Amblyopia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding and personnel are lack.
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1307011930
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Amblyopia
Keywords: amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 4-hour AmblyZ glasses (Experimental): 4-hour AmblyZ glasses for moderate amblyopia
  Interventions: Device: 4-hour AmblyZ glasses
- 2-hour eye patching (Active Comparator): 2-hour eye patching for moderate amblyopia
  Interventions: Device: 2-hour patching
- 12-hour AmblyZ glasses (Experimental): 12-hour AmblyZ glasses for severe amblyopia
  Interventions: Device: 12-hour AmblyZ glasses
- 6-hour eye patching (Active Comparator): 6-hour eye patching for severe amblyopia
  Interventions: Device: 6-hour patching

INTERVENTIONS:
Device: 4-hour AmblyZ glasses — 4-hour AmblyZ glasses for moderate amblyopia
  Arms: 4-hour AmblyZ glasses
Device: 12-hour AmblyZ glasses — 12-hour AmblyZ glasses for severe amblyopia
  Arms: 12-hour AmblyZ glasses
Device: 2-hour patching — 2-hour patching for moderate amblyopia
  Arms: 2-hour eye patching
Device: 6-hour patching — 6-hour patching for severe amblyopia
  Arms: 6-hour eye patching

SUMMARY:
Electronic eyeglasses, Amblyz™glasses, are a new medical device designed to treat amblyopia, which intermittently become opaque and provide effective occlusion for 50% of the time they are worn. A non-randomized study reported that Amblyz glasses yield an improvement in the amblyopic eye and offer an alternative effective treatment. We are unaware of any randomized clinical trial reports of response to AmblyzTM glasses treatment of amblyopia.

Our hypothesis: Amblyz™glasses can improve visual acuity of the amblyopic eye as effective as traditional patching treatment.

The primary objective is to determine if AmblyzTM equally treats moderate amblyopia as the standard 2-hour patching treatment and AmblyzTM equally treats severe amblyopia as the standard 6-hour patching treatment.

This study is designed to evaluate the effectiveness of a novel amblyopia treatment, AmblyzTM glasses, in treating amblyopia.

Moderate amblyopia: Children ages 3 to <8 years with visual acuity of 20/40 to 20/80 in the amblyopic eye will be enrolled and randomized into two groups: 4-hour AmblyzTM glasses treatment group and standard 2-hour patching control group.

Severe amblyopia: Children ages 3 to <8 years with visual acuity of 20/100 to 20/400 in the amblyopic eye will be enrolled and randomized into two groups: 12-hour AmblyzTM glasses treatment group and standard 6-hour patching control group.

ELIGIBILITY:
Inclusion Criteria:

* Both genders and all races are eligible to this study.
* Age 3 to 8 years
* Amblyopia associated with strabismus, anisometropia, or both
* Visual acuity in the amblyopic eye between 20/40 and 20/80 inclusive
* Visual acuity in the sound eye 20/40 or better and inter-eye acuity difference >3 logarithm of the minimum angle of resolution (logMAR) lines
* Wearing of optimal spectacle correction for a minimum of 4 weeks at the time of enrollment.

Exclusion Criteria:

• No amblyopia treatment before enrollment.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Wang J, Neely DE, Galli J, Schliesser J, Graves A, Damarjian TG, Kovarik J, Bowsher J, Smith HA, Donaldson D, Haider KM, Roberts GJ, Sprunger DT, Plager DA. A pilot randomized clinical trial of intermittent occlusion therapy liquid crystal glasses versus traditional patching for treatment of moderate unilateral amblyopia. J AAPOS. 2016 Aug;20(4):326-31. doi: 10.1016/j.jaapos.2016.05.014. Epub 2016 Jul 12. PMID 27418249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 patients were consented; 45 entered the trial, with 27 assigned to the IO therapy group and 18 to the patching group.
Pre-assignment Details: 49 patients were consented; 4 patients were not qualified.
  45 entered the trial, with 27 assigned to the IO therapy group and 18 to the patching group
Period: Overall Study
Arm/Group | 4-hour AmblyZ Glasses | 2-hour Eye Patching | 12-hour AmblyZ Glasses | 6-hour Eye Patching
Started | 27 | 18 | 0 | 0
Completed | 19 | 15 | 0 | 0
Not Completed | 8 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-hour AmblyZ Glasses | 2-hour Eye Patching | 12-hour AmblyZ Glasses | 6-hour Eye Patching | Total
Number analyzed (Participants) | 19 | 15 | 0 | 0 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 15 |  |  | 34
  Between 18 and 65 years | 0 | 0 |  |  | 0
  >=65 years | 0 | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: year old] | 5.7 (1.5) | 5.9 (0.9) |  |  | 5.8 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 |  |  | 12
  Male | 14 | 8 |  |  | 22
Region of Enrollment [Number; unit: participants]
  United States | 19 | 15 |  |  | 34

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Change During 12 Weeks
Description: Visual acuity change during 12 weeks: the difference of visual acuity at baseline and 12 weeks.
Time Frame: 12 weeks
Population: Visual acuity change over 12 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | 4-hour AmblyZ Glasses | 2-hour Eye Patching | 12-hour AmblyZ Glasses | 6-hour Eye Patching
Number analyzed (Participants) | 19 | 15 | 0 | 0
logMAR | .15 (.12) | .15 (.11) |  |
Statistical Analysis 1: Comparison: 4-hour AmblyZ Glasses vs 2-hour Eye Patching; Test type: Non-Inferiority or Equivalence — A sample size of 12 subjects per group has been shown to be effective for estimating within-group means and variances when little prior data is available.(Julius, 2005) Based on collected data from 34 subjects and effective size difference of 0.1, we reestimate this study as a noninferiority trial with continuous outcome and power calculated as approximately 80%; p = 0.88, t-test, 1 sided

2. Other Pre Specified Outcome: Reverse Amblyopia
Description: it is defined that the strong eye of the patient decreases two logMAR lines over 3 months.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 4-hour AmblyZ Glasses | 2-hour Eye Patching | 12-hour AmblyZ Glasses | 6-hour Eye Patching
Number analyzed (Participants) | 19 | 15 | 0 | 0
Participants | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Significant Ocular Deviation Increase From the Baseline
Description: The significant ocular deviation is defined as equal or over 10 degrees of deviation more than that of the baseline.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 4-hour AmblyZ Glasses | 2-hour Eye Patching | 12-hour AmblyZ Glasses | 6-hour Eye Patching
Number analyzed (Participants) | 19 | 15 | 0 | 0
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: In addition to monitoring all Serious and non-serious adverse events, participants were specifically monitored/assessed for the following two major Other adverse events:
  1. reverse amblyopia (the fellow good eye becomes two logMAR line worse than the amblyopic eye)
  2. Significant deviation increase than baseline.
Arm/Group | 4-hour AmblyZ Glasses | 2-hour Eye Patching | 12-hour AmblyZ Glasses | 6-hour Eye Patching
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. Sample size is limited; some patients did not come for followup visit.
2. Compliance with treatment is only estimated with calendar log and many patients did not bring back report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes